CLINICAL TRIAL: NCT01510054
Title: Endometrial Luteal Phase Characteristics and Luteal Phase Support in Controlled Ovarian Stimulation Protocols With Gonadotropin Releasing Hormone (GnRH) Antagonists: Focusing on MicroRNA Identification and Expression
Brief Title: Endometrial Luteal Phase Characteristics and Luteal Phase Support in Controlled Ovarian Stimulation Protocols With GnRH Antagonists:Focusing on MicroRNA
Status: Withdrawn | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IISP 38749
Record Dates: First submitted 2011-12-22; First posted 2012-01-13 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Controlled Ovarian Stimulation
Keywords: miRNA in endometrium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — endometril tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- steroid support: Endometrial biopsies from subjects of with or without luteal phase steroid support will be compared for miRNA expression

SUMMARY:
MiRNAs are single-stranded small non-coding RNAs that act on specific mRNAs to regulate the gene expression. Studies have suggested that miRNAs influence cellular activities in the uterus, including cell differentiation and embryo implantation.

In assisted reproductive cycles, controlled ovarian stimulation (COS) results in supraphysiological steroid levels and is associated with very low luteinizing hormone concentration during the luteal phase, the peri-implantation and implantation period. Luteal phase support, administration of medication aimed at supporting the implantation process, has been a routine practice in in vitro fertilization (IVF) clinics. Luteal phase support with steroid hormone has been found to improve pregnancy rates when human menopausal gonadotropins were used in conjunction with GnRH agonists for ovarian stimulation and IVF. Reports on effect of steroid supplementation in GnRH antagonist protocols are limited.

The proposed project is an extension of our previous study on Endometrial Luteal Phase Characteristics and Luteal Phase Support in Controlled Ovarian Hyperstimulation Protocols with Gonadotropin Releasing Hormone Antagonists. The significance of this study is based on the importance of luteal phase endometrial after COS for the process of implantation. The availability of oocycte donors in assisted reproduction technology programs offers a unique opportunity to study the impact of different stimulation protocols on the quality of the luteal phase. In addition, the oocyte donor model may allow us to evaluate the impact of different luteal support protocols directly on the endometrial preparation by histological as well as biochemical markers.

Study design: Study subjects underwent ovarian stimulation according to a gonadotropin/GnRH antagonist protocol. All donors had a baseline measurement of serum follicle stimulating hormone (FSH) and estradiol levels on the second day of their menstrual cycles. Provided serum FSH levels were less than 10mIU/ml and E2 levels were less than 60pg/ml, ovarian stimulation was initiated with recombinant FSH. The daily dose was adjusted according to follicular development by serial transvaginal ultrasound and serum E2 response. A daily evening dose of ganirelix acetate was initiated on the 6th day of stimulation and continued through the day of human chorionic gonadotropin administration. When at least three follicles reached a mean diameter of 18mm, ovulation was triggered with a single dose of Human chorionic gonadotropin (hCG). Sonographically guided transvaginal oocyte retrieval was performed 34-36 hours after the hCG administration.

Thirty endometrial biopsies from oocyte donors on their COS cycles will be used for the study. Study subjects have been randomized into 4 groups. Grp 1: day of retrieval, did not receive any luteal-phase support, which serves as base line; grp2: 3, 5 and 10 days after retrieval with no luteal phase support, which serves as control; grp3: 3, 5 and 10 days after retrieval, luteal phase support with progesterone in the form of vaginal suppositories starting from the day after retrieval; grp4: daily oral dose of 2 mg 17β-estradiol in addition to the micronized progesterone. Immediately after the endometrial biopsy all specimens were stored in liquid nitrogen tanks at -196°C.

Total RNA will be isolated and microarray will be performed using an Illumina miRNA expression panel. Array results will be compiled and analyzed focusing on the following aspects: the target genes of prominent miRNAs, miRNA profile in relation to target gene pathways; miRNA expression profile in relation to endometrial dating and status; effect of luteal phase support on miRNA expression after ovarian stimulation. Minimum of 3 miRNA arrays will be run for each sample for the purpose of statistical analysis. A total of 30 arrays will be needed for all samples from all groups.

In this study, the investigators pose three questions: 1) How many and what types of miRNAs are in the endometrium during ovarian stimulation? This is to identify miRNAs and associated target genes that are relevant for endometrium receptivity; 2) Do levels of miRNA expression change during the luteal phase, or during the window of implantation? This is to examine the dynamics of miRNAs that are associated with remodeling process of endometrium; and 3) Do luteal phase support alter miRNA expression in the luteal phase? This is to investigate the steroid effect on miRNA regulation. The investigators hypothesize that many critical genes related to implantation are regulated by miRNAs. This research effort will potentially advance our knowledge of endometrial characteristics after COS and the impact of sex steroid supplementation. Overall the study should help better understand the genetic control of implantation. Completion of this study may also provide measurable scientific evidence and useful information for the management of IVF cycles.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 31 years of age female who underwent a standard screening protocol for oocyte donation, in accordance with the recommendations of the American Society for Reproductive Medicine.

Exclusion Criteria:

* Women with a body mass index exceeding 28 kg/m2,
* history of:

  * pelvic inflammatory disease,
  * sexually transmitted diseases,
  * reproductive tract pathology, or
  * other systemic diseases or conditions

Ages: 21 Years to 31 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 emdometrial biopsy from oocyte donors
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2002-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
microRNA expression in human endometrium after IVF | Up to 4 years are estimated for the study to be completed including all measures.

CONTACTS AND LOCATIONS:
Overall Officials: Yulian Zhao, Ph.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins at Green Spring Station, Lutherville, Maryland, United States